CLINICAL TRIAL: NCT00305838
Title: Use of Changes in CA 125 Doubling Time to Detect Activity of Cytostatic Agents in Women Relapsing With Ovarian Carcinoma. Study 1-Tamoxifen
Brief Title: CA 125 Levels in Treating Patients With Relapsed Advanced Ovarian Cancer, Fallopian Tube Cancer, or Primary Peritoneal Cancer Who Are Receiving Tamoxifen
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mount Vernon Cancer Centre at Mount Vernon Hospital (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000463518; CDR0000463518 (Registry Identifier: PDQ (Physician Data Query)); EU-205113; NCRN-1509; MREC-EC2003-62
Record Dates: First submitted 2006-03-21; First posted 2006-03-22 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2009-06

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; stage IIIA ovarian epithelial cancer; stage IIIB ovarian epithelial cancer; stage IIIC ovarian epithelial cancer; recurrent fallopian tube cancer; stage IIIA fallopian tube cancer; stage IIIB fallopian tube cancer; stage IIIC fallopian tube cancer; stage IV fallopian tube cancer; recurrent primary peritoneal cavity cancer; stage IIIA primary peritoneal cavity cancer; stage IIIB primary peritoneal cavity cancer; stage IIIC primary peritoneal cavity cancer; stage IV primary peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Tamoxifen

INTERVENTIONS:
Drug: tamoxifen citrate
Other: diagnostic laboratory biomarker analysis

SUMMARY:
RATIONALE: Estrogen may cause the growth of ovarian cancer cells. Hormone therapy using tamoxifen may fight ovarian cancer by blocking the use of estrogen by the tumor cells. Measuring CA 125 levels may help doctors predict a patient's response to tamoxifen and help plan the best treatment.

PURPOSE: This phase II trial is studying CA 125 levels in treating patients with relapsed advanced ovarian cancer, fallopian tube cancer, or primary peritoneal cancer who are receiving tamoxifen.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the percentage of patients with relapsed advanced ovarian carcinoma, fallopian tube carcinoma, or primary peritoneal carcinoma who have a log linear rise in CA 125 levels.
* Determine whether the log linear part of the curve is consistent enough to allow comparison of the slope before and after introduction of a new therapy.
* Compare the serial doubling time before and after commencing tamoxifen citrate treatment.
* Determine the number of patients required to detect a significant difference in CA 125 doubling time before and after starting tamoxifen citrate treatment.

OUTLINE: Patients undergo blood collection once a month to measure CA 125 levels. Once the CA 125 level goes above the upper limit of normal (ULN) or has started to rise from its nadir level (if not previously normal), CA 125 levels are measured every 2 weeks. When CA 125 levels reach 4 times the ULN or 4 times the nadir level (if not previously normal), patients begin oral tamoxifen citrate once daily for 3-6 months in the absence of disease progression or unacceptable toxicity. CA 125 levels will continue to be measured every 2 weeks during treatment.

PROJECTED ACCRUAL: A total of 200 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced ovarian carcinoma, fallopian tube carcinoma, or primary peritoneal carcinoma
* Completed therapy for first relapse

  * Had an elevated CA 125 level before starting relapse therapy with ≥ 50% fall by completion of that therapy or response according to RECIST criteria
* No significant cancer-related symptoms requiring urgent treatment

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 3 months
* Hemoglobin > 10 g/dL
* WBC > 2,500/mm^3
* Platelet count > 100,000/mm^3
* Creatinine < 2 times upper limit of normal (ULN)
* AST/ALT < 2 times ULN
* Bilirubin < 1.5 times ULN
* No evidence of significant clinical disorder or laboratory finding that would preclude study participation
* No psychiatric disorder that would preclude informed consent
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

* No other concurrent hormonal therapy, except hormone-replacement therapy
* Other concurrent medications allowed provided dose is stable

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2004-03; Primary Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who have a log linear rise in CA 125 levels
Comparison of the slope before and after introduction of a new therapy in terms of consistency of the log linear part of the curve
Comparison of the serial doubling time before and after commencing tamoxifen
Number of patients required to detect a significant difference in CA 125 doubling time before and after starting tamoxifen

CONTACTS AND LOCATIONS:
Overall Officials: Gordon J.S. Rustin, MD, Study Chair — Mount Vernon Cancer Centre at Mount Vernon Hospital
Locations (24):
- United Kingdom (24):
  - Queen's Hospital, Burton-on-Trent, England
  - Chelmsford and Essex Centre, Chelmsford, England
  - Royal Derby Hospital, Derby, England
  - St. Luke's Cancer Centre at Royal Surrey County Hospital, Guildford, England
  - Ipswich Hospital, Ipswich, England
  - Airedale General Hospital, Keighley, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Liverpool Women's Hospital, Liverpool, England
  - Saint Bartholomew's Hospital, London, England
  - Clatterbridge Centre for Oncology, Merseyside, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England
  - Kings Mill Hospital, Nottinghamshire, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Wexham Park Hospital, Slough, Berkshire, England
  - Southampton General Hospital, Southampton, England
  - Great Western Hospital, Swindon, England
  - Hillingdon Hospital, Uxbridge, England
  - NHS Grampian, Aberdeen, Scotland
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - North Glasgow University Hospitals NHS Trust, Glasgow, Scotland
  - Ysbyty Gwynedd, Bangor, Wales
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales
  - Glan Clwyd Hospital, Rhyl, Denbighshire, Wales
  - Wrexham Maelor Hospital, Wrexham, Wales